CLINICAL TRIAL: NCT02279121
Title: Prospective, Randomized, Controlled Trial Evaluating the Efficacy of a Lock-therapy With a Solution of Taurolidine/Citrate (TauroLock) vs Standard Saline Solution for the Primary Prevention of Catheter-related Infections (CLI) in Adult Patients Wtih a Non-hematological Cancer Treated With Intravenous Anti-tumor Therapy
Brief Title: ATAPAC Study (TauroLock Activity in Adult Cancer Patients)
Acronym: ATAPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Collaborators: centre régional de pharmacovigilance de Nancy (Unknown); Theradial (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-01-CHRMT; 2014-A01117-40 (Registry Identifier: ID RCB)
Record Dates: First submitted 2014-10-09; First posted 2014-10-30 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Catheter-Related Infections
Keywords: central venous catheter; Taurolidine; lock-therapy
MeSH Terms: conditions — Catheter-Related Infections | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TauroLock (Experimental): solution of taurolidine-citrate
  Interventions: Device: Taurolock
- Control (Other): saline solution
  Interventions: Drug: saline solution

INTERVENTIONS:
Device: Taurolock — At the beginning of each course of IV anti-tumor treatment, a nurse removes the lock TauroLock ™ and makes rinsing the CVC. At the end of each course, she rinses again the CVC and instills TauroLock ™ solution. Patients will be followed for each treatment, according to the same rhythm of their anti-tumor treatment program up to the end of the study
  Other Names: solution of taurolidine-citrate
  Arms: TauroLock
Drug: saline solution — At the beginning of each course of IV anti-tumor treatment, a nurse makes rinsing the CVC. At the end of each course, she rinses again the CVC. Patients will be followed for each treatment, according to the same rhythm of their anti-tumor treatment program up to the end of the study
  Arms: Control

SUMMARY:
The purpose of this study is to compare the efficacy of a lock taurolidine-citrate solution vs standard saline solution for primary prevention of central venous catheter-associated bloodstream infection in adult patients treated with intra-venous therapy for a solid tumor

DETAILED DESCRIPTION:
The central venous catheter (CVC)-associated bloodstream infection (CLABSI) represent a serious and persistent health problem in cancer patients with an implantable CVC receiving an intravenous (IV) anti-tumor therapy. The CLABSI include the CVC-associated bacteremia and the negative bloodstream local or generalized infections. CLABSI significantly increase morbidity and hospital costs. They can lead also to discontinuation of IV anti-tumor treatment, a severe sepsis, a septic shock or a death. Microbial colonization and biofilm development, which are resistant to antibiotic therapy, often lead to CVC replacement. CLABSI prevention is a key measure to improve clinical outcomes, particularly in patients at high risk. For this reason, CLABSI prevention is a national priority of the healthcare program. Taurolidine [bis-(1,1-dioxoperhydro-1,2,4-thiadiazinyl-4) methane] is an antimicrobial agent which kills and inhibits a wide range of micro-organisms in vitro, including multidrug resistant bacteria. A catheter lock solution was developed containing 1.35% taurolidine and 4% citrate. Due to the anti-adhesion activity of the taurolidine and anti-thrombotic properties of the citrate, this lock solution can disrupt bacterial adhesion to the inner surface of the implantable CVC preventing the production of biofilm. This lock solution showed a substantial reduction in the formation of biofilm and bacterial colonization of the inner surface of the implantable CVC is several prospective trials.

In a study of pediatric cancers receiving IV anti-tumor treatment, the use of a lock solution of taurolidine-citrate resulted in a reduction of Gram-positive CLABSI as compared to a control group of patients treated with a standard heparin lock solution. In another study of 71 pediatric patients, taurolidine-citrate solution reduced CLABSI compared with heparin (0.3 vs 1.3 infections per 1000 catheter-days, p: 0.03). Microbial colonization was found in 25.4% of the catheters. Regarding the toxicity, 7 patients only in the taurolidine-citrate group (20%) experienced side effects, the most being nausea, vomiting and abnormal sensations of taste.

Some clinical trials have also demonstrated the efficacy of taurolidine-citrate in terms of CLABSI reduction in patients on home total parenteral nutrition and in hemodialysis patients.

According to the French guidelines, an anti-bacterial lock therapy (preferably taurolidine) may be used as prevention in patients at increased risk of serious CLABSI complications. However, the effectiveness of the lock taurolidine-citrate solution for adult patients with solid tumors receiving an anti-tumor treatment via a totally implantable CVC is actually unknown and it remains to be assessed.

PRIMARY OBJECTIVE

- To compare the efficacy of a lock taurolidine-citrate solution vs standard saline solution for primary prevention of CLABSI in adult patients treated with IV anti-tumor therapy for a solid tumor.

SECONDARY OBJECTIVES

* To compare the impact of CLABSI in the 2 groups in terms of days of hospitalisation, delay of IV anti-tumoral treatment, costs of CVC removal and CLABSI-management
* To evaluate the adverse effects of the lock taurolidine-citrate solution in adult patients receiving an IV anti-tumor therapy for solid tumor PRIMARY ENDPOINT: Incidence rates of CLABSI per 1000 catheter-days

SECONDARY ENDPOINTS

* Days of CLABSI-related hospitalisation
* Anti-tumor treatment CLABSI-related delay
* Total CVC-removal for CLABSI
* Costs associated with the CLABSI management in the perspective of health insurance
* Evaluation of the taurolidine-citrate solution-related adverse effects

METHODOLOGY

* Single-center prospective, randomized, open-label, controlled, clinical phase IV trial
* 1:1 randomization

Stratification:

* Metastatic vs (neo) adjuvant
* Age ≤ 70 years vs > 70 years

PROCEDURES During a standard clinical visit for IV anti-tumor treatment administration, the investigator informs the patient of the study procedures and check the eligibility criteria. At the beginning of the next cure, he collects his informed consent and performs randomisation. The patient is then included in the TauroLock ™ or saline arm.

At the beginning of each course, a nurse removes the lock TauroLock ™ and / or makes rinsing the CVC. At the end of each course, she rinses again the CVC and instills TauroLock ™ solution for patients in the TauroLock ™ arm. Patients will be followed for each treatment, according to the same rhythm of their anti-tumor treatment program up to the end of the study: the end of the IV anti-tumor treatment, the CVC removal for mechanical reasons or a CLABSI.

A follow-up visit will be performed 7-30 days after the study end.

PATIENTS NUMBER Based on surveillance data of nosocomial infections at our institution, the incidence of CLABSI in the control group is expected to about 3 per 1000 catheter-days.

Assuming that the use of TauroLock ™ will reduce at least this rate by three (expected 1 per 1000 in the treated group rate), which is consistent with literature data, 9785 days must be followed in each group (α and β risk at 5% and 10%, respectively).

Considering a mean follow-up of 4 months, we need for 81 patients pour any treatment group, 162 patients for the 2 groups.

TRIAL TIME

Duration of the inclusion period:

- 6 months

Duration of participation for each patient:

- Duration of IV anti-tumor treatment + 1 month of follow-up

STATISTICAL ANALYSIS Verification of the homogeneity of the groups for major confounding factors: WHO performance status, indication for anti-tumor treatment (metastatic vs (neo)-adjuvant cancer), age, duration of follow-up, type of anti-tumor treatment (weekly, every 15 or 21 days) and type of hospitalisation (full vs day-hospital). Qualitative variables will be compared between the 2 groups by Chi-square test or Fisher exact test if the normality conditions are not met. Quantitative variables are compared by Student's t test or non parametric Wilcoxon test if the normality conditions are not met.

Primary endpoint: the incidence of CLABSI will be compared between groups by a logistic regression test with adjustment for stratification and confounding factors, if necessary.

Secondary endpoints: the qualitative criteria will be compared between the 2 groups by Chi-square test or Fisher exact test if the conditions of normality are not met. The quantitative criteria will be compared by Student's t test or non parametric Wilcoxon test if the conditions of normality are not met.

The α risk is set at 5%.

EXPECTED BENEFITS The expected benefits are a direct reduction of CLABSI for adult cancer patients receiving IV anti-tumor treatment via a CVC leading to a direct reduction of morbidity and mortality. In addition, a better control of CLABSI should allow a cost savings. A literature review by the Centers for Disease Control and Prevention (Atlanta, USA) estimated between $ 29,156 and 7288 the cost of CLABSI. Similarly, a report by the Institute for Research and Documentation in Health Economics (IRDES), based on the PMSI (Program of medicalization of information systems) data, estimated that CLABSI entailed an additional cost of € 10,950 (+ / - 1690) and a extending of the hospitalisation of 14.7 days (+ / - 1.84). Finally, a reduction of the CLABSI should globally lead to a less use of antibiotics and to a consequently reduced probability of resistant organisms selection.

QUALITY ASSURANCE PLAN Data will be recorded in a paper case report form from medical records.

The accuracy and completeness of data will be monitored by a study coordinator :

* 100% inform consent, eligibility criteria and safety data
* 20% data recorded in CRF (case report form) Data will be registered in Microsoft Office ACCESS 2003 Base. It's a single-center study so thre're no special procedures to address registry operations and analysis activities. Safety data like reporting for adverse event will be made by fax with The CRPV (centre régional de pharmacovogilance de Nancy).

The security of the data transfer is assured by the french "Méthodologie de Référence MR001" (Comission Nationale Informatique et Liberté).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Performance Index (WHO score) ≤ 2
* Patient with a solid cancer receiving an IV anti-tumor treatment
* Presence of a totally implantable CVC
* Anti-tumoral therapy administered by a totally implantable CVC
* Metastatic and / or (neo) adjuvant treatment
* Full hospitalised and / or day-hospital patients
* Informed written consent
* Social Health security insurance

Exclusion Criteria:

* Hematological cancer patients
* HIV-positive patients and/ or patients receiving an active immunosuppressive therapy
* Patients presenting a febrile episode within 4 days prior to randomisation
* Patients with neutropenia grade ≥ 2 (ANC ≤ 1000/mm3) on a blood testing older than 7 days
* Patients on IV antibiotic therapy
* Patients on total and / or peripheral parental nutrition
* Patients with a previous CLABSI history
* Allergy to citrate or taurolidine
* Patients who are not able to give an informed consent
* Patients under guardianship
* Patients under judicial protection
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
central venous catheter-associated bloodstream infection (CLABSI) | during the IV anti-tumor treatment + 1 month of follow-up = 5 months on average and for up to 11 months
  incidence rates of CLABSI per 1000 catheter-days

SECONDARY OUTCOMES:
days of CLABSI-related hospitalisation | during the IV anti-tumor treatment + 1 month of follow-up = 5 months on average and for up to 11 months
Anti-tumor treatment CLABSI-related delay | during the IV anti-tumor treatment + 1 month of follow-up = 5 months on average and for up to 11 months
Total CVC removal for CLABSI | during the IV anti-tumor treatment + 1 month of follow-up = 5 months on average and for up to 11 months
Costs associated with the CLABSI management in the perspective of health insurance | during the IV anti-tumor treatment + 1 month of follow-up = 5 months on average and for up to 11 months
Evaluation of the taurolidine-citrate solution-related adverse effects | during the IV anti-tumor treatment + 1 month of follow-up = 5 months on average and for up to 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele LONGO, MD, Principal Investigator — CHR Metz Thionville
Locations (1):
- Chr Metz Thionville, Metz, France

REFERENCES:
- [Background] Quarello F, Forneris G. Prevention of hemodialysis catheter-related bloodstream infection using an antimicrobial lock. Blood Purif. 2002;20(1):87-92. doi: 10.1159/000046990. PMID 11803164
- [Background] Allon M. Prophylaxis against dialysis catheter-related bacteremia with a novel antimicrobial lock solution. Clin Infect Dis. 2003 Jun 15;36(12):1539-44. doi: 10.1086/375234. Epub 2003 Jun 6. PMID 12802753
- [Background] Betjes MG, van Agteren M. Prevention of dialysis catheter-related sepsis with a citrate-taurolidine-containing lock solution. Nephrol Dial Transplant. 2004 Jun;19(6):1546-51. doi: 10.1093/ndt/gfh014. Epub 2004 Feb 19. PMID 14993498
- [Background] Mandolfo S, Borlandelli S, Elli A. Catheter lock solutions: it's time for a change. J Vasc Access. 2006 Jul-Sep;7(3):99-102. doi: 10.1177/112972980600700302. PMID 17019660
- [Background] Taylor C, Cahill J, Gerrish M, Little J. A new haemodialysis catheter-locking agent reduces infections in haemodialysis patients. J Ren Care. 2008 Sep;34(3):116-20. doi: 10.1111/j.1755-6686.2008.00027.x. PMID 18786077
- [Background] Solomon LR, Cheesbrough JS, Ebah L, Al-Sayed T, Heap M, Millband N, Waterhouse D, Mitra S, Curry A, Saxena R, Bhat R, Schulz M, Diggle P. A randomized double-blind controlled trial of taurolidine-citrate catheter locks for the prevention of bacteremia in patients treated with hemodialysis. Am J Kidney Dis. 2010 Jun;55(6):1060-8. doi: 10.1053/j.ajkd.2009.11.025. Epub 2010 Mar 6. PMID 20207458
- [Background] Filiopoulos V, Hadjiyannakos D, Koutis I, Trompouki S, Micha T, Lazarou D, Vlassopoulos D. Approaches to prolong the use of uncuffed hemodialysis catheters: results of a randomized trial. Am J Nephrol. 2011;33(3):260-8. doi: 10.1159/000324685. Epub 2011 Mar 2. PMID 21372561
- [Background] Solomon LR, Cheesbrough JS, Bhargava R, Mitsides N, Heap M, Green G, Diggle P. Observational study of need for thrombolytic therapy and incidence of bacteremia using taurolidine-citrate-heparin, taurolidine-citrate and heparin catheter locks in patients treated with hemodialysis. Semin Dial. 2012 Mar-Apr;25(2):233-8. doi: 10.1111/j.1525-139X.2011.00951.x. Epub 2011 Sep 15. PMID 21916999
- [Background] Zhao Y, Li Z, Zhang L, Yang J, Yang Y, Tang Y, Fu P. Citrate versus heparin lock for hemodialysis catheters: a systematic review and meta-analysis of randomized controlled trials. Am J Kidney Dis. 2014 Mar;63(3):479-90. doi: 10.1053/j.ajkd.2013.08.016. Epub 2013 Oct 11. PMID 24125729
- [Background] Toure A, Lauverjat M, Peraldi C, Boncompain-Gerard M, Gelas P, Barnoud D, Chambrier C. Taurolidine lock solution in the secondary prevention of central venous catheter-associated bloodstream infection in home parenteral nutrition patients. Clin Nutr. 2012 Aug;31(4):567-70. doi: 10.1016/j.clnu.2012.01.001. Epub 2012 Jan 28. PMID 22285029
- [Background] Lebeaux D, Larroque B, Gellen-Dautremer J, Leflon-Guibout V, Dreyer C, Bialek S, Froissart A, Hentic O, Tessier C, Ruimy R, Pelletier AL, Crestani B, Fournier M, Papo T, Barry B, Zarrouk V, Fantin B. Clinical outcome after a totally implantable venous access port-related infection in cancer patients: a prospective study and review of the literature. Medicine (Baltimore). 2012 Nov;91(6):309-318. doi: 10.1097/MD.0b013e318275ffe1. PMID 23117849
- [Background] Zwiech R, Adelt M, Chrul S. A Taurolidine-Citrate-Heparin Lock Solution Effectively Eradicates Pathogens From the Catheter Biofilm in Hemodialysis Patients. Am J Ther. 2016 Mar-Apr;23(2):e363-8. doi: 10.1097/MJT.0b013e31828d4610. PMID 23665885
- [Background] Shah CB, Mittelman MW, Costerton JW, Parenteau S, Pelak M, Arsenault R, Mermel LA. Antimicrobial activity of a novel catheter lock solution. Antimicrob Agents Chemother. 2002 Jun;46(6):1674-9. doi: 10.1128/AAC.46.6.1674-1679.2002. PMID 12019075
- [Background] Torres-Viera C, Thauvin-Eliopoulos C, Souli M, DeGirolami P, Farris MG, Wennersten CB, Sofia RD, Eliopoulos GM. Activities of taurolidine in vitro and in experimental enterococcal endocarditis. Antimicrob Agents Chemother. 2000 Jun;44(6):1720-4. doi: 10.1128/AAC.44.6.1720-1724.2000. PMID 10817739
- [Background] Simon A, Ammann RA, Wiszniewsky G, Bode U, Fleischhack G, Besuden MM. Taurolidine-citrate lock solution (TauroLock) significantly reduces CVAD-associated grampositive infections in pediatric cancer patients. BMC Infect Dis. 2008 Jul 29;8:102. doi: 10.1186/1471-2334-8-102. PMID 18664278
- [Background] Dumichen MJ, Seeger K, Lode HN, Kuhl JS, Ebell W, Degenhardt P, Singer M, Geffers C, Querfeld U. Randomized controlled trial of taurolidine citrate versus heparin as catheter lock solution in paediatric patients with haematological malignancies. J Hosp Infect. 2012 Apr;80(4):304-9. doi: 10.1016/j.jhin.2012.01.003. Epub 2012 Feb 18. PMID 22342714
- [Background] Klek S, Szczepanek K, Hermanowicz A, Galas A. Taurolidine lock in home parenteral nutrition in adults: results from an open-label randomized controlled clinical trial. JPEN J Parenter Enteral Nutr. 2015 Mar;39(3):331-5. doi: 10.1177/0148607114525804. Epub 2014 Mar 6. PMID 24604029
- [Background] Al-Amin AH, Sarveswaran J, Wood JM, Burke DA, Donnellan CF. Efficacy of taurolidine on the prevention of catheter-related bloodstream infections in patients on home parenteral nutrition. J Vasc Access. 2013 Oct-Dec;14(4):379-82. doi: 10.5301/jva.5000168. Epub 2013 Jul 1. PMID 23817948
- See also: Prévention des infections associées aux chambres à cathéter implantables pour accès veineux. Recommandations professionnelles par consensus formalisé d'experts. Mars 2012 — http://www.sf2h.net/
- See also: Nestrigue, C., Or, Z. Surcoût des événements indésirables associés aux soins à l'hôpital. Premières estimations à partir de neuf indicateurs de sécurité des patients. Document de Travail IRDES n°44. Février 2012 — http://www.irdes.fr/EspaceRecherche/DocumentsDeTravail/DT44EstimationSurcoutsEvenementsIndesSoinsHopitalFrance.pdf
- See also: Ministère de la santé, de la jeunesse et des sports DGS/DHOS, CTINILS. Définition des infections associées aux soins (mai 2007) — http://www.sante.gouv.fr/IMG/pdf/rapport_vcourte.pdf